CLINICAL TRIAL: NCT03585426
Title: Vancomycin in the Target Site Treatment of Intracranial Infection : a New Strategy for PK/PD Treatment
Brief Title: Vancomycin in the Target Site Treatment of Intracranial Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJYY-LL-FJ-045
Record Dates: First submitted 2018-07-01; First posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-06

CONDITIONS: Vancomycin
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vancomycin 1g q12h (Experimental)
  Interventions: Drug: Vancomycin
- Vancomycin 1g q8h (Experimental)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Vancomycin, a novel intravenously administered glycylcycline antibiotic, currently plays a key role in the management of complicated multi-organism infections.

SUMMARY:
Vancomycin, a novel intravenously administered antibiotic, currently plays a key role in the management of complicated multi-organism infections. However,current LC-MS/MS methods briefly describe parameters and the only reported internal standard was sometimes difficult to obtain. In our study,an updated LC-MS/MS method for the quantitative analysis of vancomycin in human serum was developed.

ELIGIBILITY:
Inclusion Criteria:

In ICU; ventricle drainage was carried out; renal function is normal, namely creatinine clearance rate is >60ml/min;

Exclusion Criteria:

women in pregnancy or lactation;in patients with renal insufficiency, the creatinine clearance rate (Clcr) is less than 60ml/min.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Vancomycin concentration change in serum and cerebrospinal fluid | 0.5h, 1h, 1.5h, 3h, 5h, 7h, 9h, and 12h after treatment
  Quantitative analysis of vancomycin in serum and cerebrospinal fluid after treatment by an updated LC-MS/MS method.

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Jia, Dr., Study Director — The First Affiliated Hospital, the Fourth Military Medical University